CLINICAL TRIAL: NCT00650078
Title: A Randomized Multi-Center, Double-Blind, Placebo-Controlled Study of a New Modified-Release Tablet Formulation of Prednisone (Lodotra®) in Patients With Rheumatoid Arthritis
Brief Title: Study to Assess the Safety and Efficacy of Modified-Release Prednisone (Lodotra®) Therapy in Patients With Active Rheumatoid Arthritis
Acronym: CAPRA-2
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NP01-007; EudraCT-Number: 2007-003508-36
Record Dates: First submitted 2008-03-28; First posted 2008-04-01 (Estimated); Results first posted 2012-12-13 (Estimated); Last update posted 2024-12-18 (Actual); Status verified 2024-11

CONDITIONS: Rheumatoid Arthritis
Keywords: Signs and Symptoms; Autoimmune Diseases; Joint Diseases; Arthritis; Connective Tissue Diseases; Arthritis, Rheumatoid; Rheumatic Diseases; Predniso(lo)ne
MeSH Terms: conditions — Arthritis, Rheumatoid; Signs and Symptoms; Autoimmune Diseases; Joint Diseases; Arthritis; Connective Tissue Diseases; Rheumatic Diseases

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- NP01 (Experimental): Modified Release (MR) prednisone 5 mg
  Interventions: Drug: MR prednisone
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: MR prednisone — 1 x 5 mg daily
  Arms: NP01
Drug: Placebo — 1x daily
  Arms: Placebo

SUMMARY:
The purpose of the study is to compare the safety and efficacy, with regards to the signs and symptoms, of MR prednisone (Lodotra®) versus placebo in combination with standard Disease Modifying Anti-Rheumatic Drug (DMARD) treatment in patients with active rheumatoid arthritis.

DETAILED DESCRIPTION:
Study with completed results acquired from Horizon in 2024.

ELIGIBILITY:
Inclusion Criteria:

* Documented history of RA in agreement with ACR criteria
* DMARD treatment for RA greater than or equal to 6 months, with a stable dose greater than or equal to 6 weeks prior to screening visit
* Duration of morning stiffness greater than or equal to 45 minutes
* greater than or equal to 4 swollen joints (out of 28)
* greater than or equal to 4 tender joints (out of 28)

Exclusion Criteria:

* Suffering from another disease, which requires glucocorticoid treatment during the study period
* Synovectomy within 4 months prior to study start
* Use of glucocorticoids:

  * Continued use of systemic glucocorticoids within 4 weeks prior to screening visit
  * Intermittent use of glucocorticoids within 2 weeks prior to screening visit.
  * Joint injections within 6 weeks prior to screening visit
  * Topical glucocorticoids must be stopped at screening visit
* Use of biologicals such as: tumor necrosis factor α (TNFα) inhibitors and other compounds within 5 serum half lives prior to screening visit
* Pregnancy or nursing

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 350 (Actual)
Dates: Start 2008-03; Primary Completion 2009-05 (Actual); Study Completion 2009-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (52):
- United States (28):
  - Rheumatology Associates of N. AL, P.C., Huntsville, Alabama
  - ArthoCare, Arthritis Care & Research, P.C., Phoenix, Arizona
  - The National Institute of Clinical Research, Los Angeles, California
  - University of California, Los Angeles, Los Angeles, California
  - Blue Hill Medical Group, Pacific Palisades, California
  - San Diego Arthritis Medical Clinic, San Diego, California
  - Boling Clinical Trials, Upland, California
  - Lynn Institute of the Rockies, Colorado Springs, Colorado
  - Front Range Clinical Research, Wheat Ridge, Colorado
  - Arthritis Center, Palm Harbor, Florida
  - West Broward Rheumatology Associates, Inc., Tamarac, Florida
  - Southwest Florida Clinical Research Center, Tampa, Florida
  - Tampa Medical Group, PA, Tampa, Florida
  - Geodyssey Research, LLC, Vero Beach, Florida
  - The Arthritis Center, Springfield, Illinois
  - Center for Arthritis and Osteoporosis, Elizabethtown, Kentucky
  - Phase III Clinical Research, Fall River, Massachusetts
  - Montana Health Research Institute, Inc., Billings, Montana
  - Arthritis Center of Reno, Reno, Nevada
  - Arthritis Associates, Belmont, North Carolina
  - Clinical Research Source, Perrysburg, Ohio
  - Health Resources of Oklahoma, Oklahoma City, Oklahoma
  - DeGarmo Institute of Medical Research, Greer, South Carolina
  - Carolina Center for Rheumatology & Arthritis Care, Rock Hill, South Carolina
  - SCRI-Marker, Memphis, Tennessee
  - Radiant Research of San Antonio Northeast, San Antonio, Texas
  - Arthritis & Osteoporosis Cntr. Of S. TX, San Antonio, Texas
  - Northwest Clinical Research Center, Bellevue, Washington
- Clinical Research and Arthritis Centre, Windsor, Ontario, Canada
- Germany (4):
  - Kerckhoff-Klinik, Bad Nauheim
  - Charité Campus Mitte, Dept. of Rheumatology and Clinical Immunology, Berlin
  - Schlosspark-Klinik, Berlin
  - Praxiszentrum, St.-Bonifatius-Straße, München
- Hungary (8):
  - Budai Irgalmasrendi Kórház, Budapest
  - Debreceni Egyetem, III. Belgyógyászati Klinika, Reumatológiai Tanszék, Debrecen
  - Kenézy Gyula Kórház-Rendelőintézet, Reumatológiai Osztály, Debrecen
  - Bács-Kiskun Megyei Kórház, Reumatológiai Osztály, Kecskemét
  - Kiskunhalasi Semmelweis Kórház Kht., Reumatológiai Osztály, Kiskunhalas
  - Pécsi Tudományegyetem, Immunológiai és Reumatológiai Klinika, Pécs
  - MÁV Kórház Szolnok, Reumatológiai Osztály, Szolnok
  - Markusovszky Kórház, Reumatológiai Osztály Szombathely, Szombathely
- Poland (8):
  - Centrum Miriada, Prywatny Gabinet Specjalistyczny Prof. Dr. Stanisława Sierakowskiego, Bialystok
  - NZOZ Centrum Medyczne Artur Racewicz, Bialystok
  - Samodzielny Publiczny Szpital Kliniczny Nr 4 w Lublinie, Klinika Reumatologii i Ukladowych Chorób Tkanki Lacznej, Lublin
  - Zaklad Opieki Zdrowotnej, Poznan - Stare Miastro, Szpital im. Józefa Strusia, Oddzial Reumatologii i Osteoporozy, Poznan
  - Wojewódzki Zespol Reumatologiczny im. Dr Jadwigi Titz-Kosko w Sopocie, Sopot
  - NZOZ "Nasz Lekarz" Praktyka Grupowa Lekarzy Rodzinnych z Przychodnia Specjalistyczna, Torun
  - Centrum Leczenia Chorób Cywilizacyjnych, Warsaw
  - Akademicki Szpital Kliniczny im. Jana Mikulicza-Radeckiego we Wroclawiu, Wroclaw
- United Kingdom (3):
  - University of Bristol, Academic Rheumatology Unit, Bristol
  - Northern Lincolnshire and Goole Hospitals NHS Foundation Trust, Diana Princess of Wales Hospital, Lincolnshire
  - Arrowe Park Hospital, Metropolitan Borough of Wirral

REFERENCES:
- [Derived] Alten R, Grahn A, Holt RJ, Rice P, Buttgereit F. Delayed-release prednisone improves fatigue and health-related quality of life: findings from the CAPRA-2 double-blind randomised study in rheumatoid arthritis. RMD Open. 2015 Aug 13;1(1):e000134. doi: 10.1136/rmdopen-2015-000134. eCollection 2015. PMID 26535146
- [Derived] Buttgereit F, Mehta D, Kirwan J, Szechinski J, Boers M, Alten RE, Supronik J, Szombati I, Romer U, Witte S, Saag KG. Low-dose prednisone chronotherapy for rheumatoid arthritis: a randomised clinical trial (CAPRA-2). Ann Rheum Dis. 2013 Feb;72(2):204-10. doi: 10.1136/annrheumdis-2011-201067. Epub 2012 May 5. PMID 22562974

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Approximately 350 patients were to be enrolled (at screening, Visit 0), with a minimum of 6 and a maximum of 28 patients at each center. It was planned to randomize (at Visit 1) a total of 294 patients in 50-55 centers in North America and Europe (Germany, Hungary, Poland and UK). First patient enrolled March, 2008; last patient contact May, 2009.
Pre-assignment Details: The study consisted of a 1 week screening phase followed by a 12 week double blind treatment phase. In addition to their standard RA medication, patients received placebo during the 1 week screening phase. The purpose of the screening phase was to establish the patient's compliance with study medication and completion of diary entries.
Period: Overall Study
Arm/Group | NP01 | Placebo
Started | 231 | 119
Completed | 217 | 106
Not Completed | 14 | 13

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | NP01 | Placebo | Total
Number analyzed (Participants) | 231 | 119 | 350
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 186 | 95 | 281
  >=65 years | 45 | 24 | 69
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.1 (9.89) | 57.5 (9.55) | 57.2 (9.76)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 192 | 102 | 294
  Male | 39 | 17 | 56
Region of Enrollment [Number; unit: participants]
  United States | 48 | 27 | 75
  Hungary | 67 | 35 | 102
  Canada | 8 | 5 | 13
  Poland | 98 | 47 | 145
  Germany | 1 | 2 | 3
  United Kingdom | 9 | 3 | 12

OUTCOME MEASURES:

1. Primary Outcome: ACR 20 Response Rate at Visit 4
Description: Responders were defined as patients whose improvement from baseline to Visit 4 (Week 12) fulfilled all 3 of the following criteria:
  * > 20% reduction in the tender joint count (0-28)
  * > 20% reduction in the swollen joint count (0-28)
  * > 20% reduction in 3 out of the 5 following additional measures:
    * Patient's assessment of pain
    * Patient's global assessment of disease activity
    * Physician's global assessment of disease activity
    * Functional Disability Index of the Health Assessment Questionnaire
    * C-reactive protein or erythrocyte sedimentation rate
Time Frame: Week 12
Population: Modified Intention to Treat (mITT) efficacy population included all patients who were randomized and received at least 1 dose of study medication. Patients were analyzed according to the treatment to which they were intended to be randomized. All missing values were imputed as non-responders.
Measure: Number; unit: participants
Arm/Group | NP01 | Placebo
Number analyzed (Participants) | 231 | 119
participants | 108 | 34
Statistical Analysis 1: Comparison: NP01 vs Placebo; Test type: Superiority or Other; p = 0.0010, Regression, Logistic — The p-value was based on logistic regression with treatment, geographic region, gender, and median age class as factors; Odds Ratio (OR) = 2.25, 95% CI 2-sided [1.39 to 3.64]

2. Secondary Outcome: Relative Reduction of Morning Stiffness
Description: Data for the duration of morning stiffness were obtained from patient diaries. Duration of morning stiffness was the difference between the time of resolution of morning stiffness and the time of wake-up. Duration of morning stiffness is the average of the morning stiffness duration (minutes) over the last 7 days prior to visit day (including day of visit). If more than 4 assessments were missing, then the duration was set to missing. Baseline was the value recorded at Week -1 (Visit 0).
Time Frame: Week 12
Population: Modified Intention to Treat (mITT) efficacy population included all patients who were randomized and received at least 1 dose of study medication. Patients were analyzed according to the treatment to which they were intended to be randomized. Excludes those participants with missing data. Analysis used last observation carried forward imputation.
Measure: Median (95% Confidence Interval); unit: Relative Change from Baseline (%)
Arm/Group | NP01 | Placebo
Number analyzed (Participants) | 216 | 107
Relative Change from Baseline (%) | -55.22 (63.583) [-69.7 to -47.9] | -34.62 (67.018) [-43.0 to -19.3]
Statistical Analysis 1: Comparison: NP01 vs Placebo; Test type: Superiority or Other; p = 0.0015, Hodges-Lehman method — Wilcoxon Rank Sum Test p-value; The difference between the treatment groups was assessed using the median and the 95% CI of the median computed using the Hodges Lehmann method; Median Difference (Final Values) = -19.6, 95% CI 2-sided [-31.7 to -6.1]

ADVERSE EVENTS:
Time Frame: Initiation of double blind treatment until end of treatment or 30 days after last study drug administration, whicever occurred later
Arm/Group | NP01 | Placebo
Serious Adverse Events (participants affected / at risk) | 1/231 | 2/119
Other Adverse Events (participants affected / at risk) | 69/231 | 49/119
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | NP01 (N=231) | Placebo (N=119)
myocardial ischaemia (Cardiac disorders) | 0 (0) | 1 (1)
chest discomfort (General disorders) | 1 (1) | 0 (0)
palpitations (Cardiac disorders) | 1 (1) | 0 (0)
cytology abnormal (Investigations) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | NP01 (N=231) | Placebo (N=119)
arthralgia (Musculoskeletal and connective tissue disorders) | 24 | 24
rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 15 | 11 — Includes rheumatoid arthritis aggravated and rheumatoid arthritis flare-up(MedDRA lowest level term)
nasopharyngitis (Infections and infestations) | 11 | 4
headache (Nervous system disorders) | 9 | 5
bronchitis (Infections and infestations) | 3 | 5
hypertension (Vascular disorders) | 5 | 1
rash (Skin and subcutaneous tissue disorders) | 4 | 1
diarrhea (Gastrointestinal disorders) | 4 | 1
back pain (Musculoskeletal and connective tissue disorders) | 3 | 1
hematuria (Renal and urinary disorders) | 1 | 3
vomiting (Gastrointestinal disorders) | 3 | 1
oedema peripheral (General disorders) | 2 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The first publication shall be the presentation of a joint, multicenter publication of the Study results. If such a multicenter publication is not submitted within 24 months after conclusion of the Study at all sites, INSTITUTION/INVESTIGATOR may publish the results from the INSTITUTION'S site individually, provided that it is submitted to SPONSOR for review and comment 60 days prior to submission for publication.